CLINICAL TRIAL: NCT03471910
Title: Clinical Non-inferiority Study Between Diosmin 600 mg Tablets and Diosmin 900 mg + Hesperidin 100 mg Tablets in Symptomatic Chronic Venous Insufficiency After 6 Months of Treatment: Single-blind, Randomized, Parallel Group Study
Brief Title: Clinical Non-inferiority Study Between Diosmin 600mg & Diosmin + Hesperidin in Symptomatic Chronic Venous Insufficiency
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundação Educacional Serra dos Órgãos (Other)
Responsible Party: Principal Investigator, Carlos Pereira Nunes, Professor of Internal Medicine, Fundação Educacional Serra dos Órgãos
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DIVC-01-12-17
Record Dates: First submitted 2018-02-27; First posted 2018-03-21 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Venous Insufficiency
Keywords: Chronic venous insufficiency; Diosmin; Hesperidin
MeSH Terms: conditions — Venous Insufficiency | interventions — Diosmin; Hesperidin

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diosmin (Experimental): Diosmin 600mg, one tablet once daily
  Interventions: Drug: Diosmin
- Diosmin + Hesperidin (Active Comparator): Diosmin 900mg + Hesperidin 100mg, one tablet once daily
  Interventions: Drug: Diosmin / Hesperidin

INTERVENTIONS:
Drug: Diosmin — Diosmin 600mg tablet, once daily
  Arms: Diosmin
Drug: Diosmin / Hesperidin — Diosmin 900 mg / Hesperidin 100mg tablet, once daily
  Arms: Diosmin + Hesperidin

SUMMARY:
Clinical non-inferiority study between Diosmin 600 mg tablets and Diosmin 900 mg + Hesperidin 100 mg tablets in symptomatic chronic venous insufficiency after 6 months of treatment. Prospective, single-blind, randomized study in parallel groups (total patient population 120, 60 subjects per treatment group), with a total of 4 clinical assessment at months 0, 2, 4, and 6 of treatment.

DETAILED DESCRIPTION:
The primary study objective is to demonstrate the clinical non inferiority of efficacy between Diosmin 600 mg tablets versus combination Diosmin 900 mg + Hesperidin 100 mg tablets in improving lower limb symptoms assessed by a 100 mm visual analogue scale (VAS) over 6 months among adult patients presenting chronic venous insufficiency of the lower limbs.

The secondary study objectives are to compare between Diosmin 600 mg tablets and combination Diosmin 900 mg + Hesperidin 100 mg tablets in terms of:

* The oral acceptability,
* The tolerability,
* The global patient's satisfaction,
* The global physician's satisfaction.

Clinical assessments will take place at the study center during the study visits at M0, M2, M4 and M6 including:

* Efficacy on venous symptoms : The VAS of 100 mm is rated by the patient from "0" = Absence of venous symptoms up to "100" = Maximal intensity of the venous symptoms. The VAS is completed by the patient at the investigator's office. This VAS globally assesses the venous symptomatology of the most symptomatic leg : Heavy legs, Painful legs, Tired legs, Sensation of swelling and/or tension in the legs).
* Acceptability : Easiness to swallow assessed by a VAS of 100 mm rated by the patient from "0" = Very easy to swallow, up to "10" = Very difficult to swallow
* Patient's global satisfaction related to the treatment efficacy : Four levels scale rated as following : bad, acceptable, good, and very good
* Investigator's global satisfaction related to the treatment efficacy : Four levels scale rated as following : bad, acceptable, good, and very good
* Tolerability (related adverse events)
* Compliance : Accountability of treatments returned by the patient

The primary endpoint will be the change between the VAS symptoms scores at M0 and M6 / end of study visit (early withdrawal). Secondary endpoints include assessments of efficacy, oral acceptability of study drug, and tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders >18 years old
* Patient presenting a C0 to C3 venous disease grade of the lower limbs, according to the clinical component of the CEAP classification,
* Clinical symptoms of chronic venous insufficiency of the lower limbs as defined by a VAS of 100 mm rated by the patient between 20 mm and 60 mm on the most symptomatic leg. The VAS is a global evaluation of the following symptoms: Heavy legs, Painful legs, Tired legs, Sensation of swelling and / or tension in the legs.
* Premenopausal female subjects not pregnant or breastfeeding, in use of reliable contraceptive
* Subject has read, understood, dated and signed the informed consent form

Exclusion Criteria:

* Treatment by compression stocking within the 2 months before inclusion
* Treatment by venotonics within the 2 months before inclusion
* Premenopausal women who are pregnant, breastfeeding or who do not wish to use contraception during the study period
* Known allergy or hypersensitivity to any component of the study drug
* Known clinically significant laboratory alterations
* CEAP levels 4, 5 & 6
* Patient with venous disease requiring surgery / chemical endovenous sclerotherapy
* Patient suffering from a painful pathology other than the venous pain in the lower limbs
* Patient with history of venous thrombosis or thromboembolic disease within the 6 months before inclusion
* Patient with alteration of general condition incompatible with his / her participation in the trial
* Patient wishing to be pregnant in the 6 following months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2018-03-20 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Change in VAS symptom scores | From pretreatment (month 0) until month 6 of the 6-month treatment period
  Change between the 100mm visual analog scale (VAS) symptoms (from 0mm [absence of venous symptoms] to 100mm [maximal intensity of venous symptoms] scores at month 0 (pretreatment) and month 6 / end of study visit (early withdrawal).

SECONDARY OUTCOMES:
Efficacy: Evolution of VAS score at each visit | From pretreatment (month 0) until month 6 of the 6-month treatment period
  Evolution of the 100mm VAS symptoms (from 0mm [absence of venous symptoms] to 100mm [maximal intensity of venous symptoms]) at each visit
Efficacy: Patient global satisfaction at each visit | From pretreatment (month 0) until month 6 of the 6-month treatment period
  Evaluation of the patient's global satisfaction at each visit on a four level scale of "bad", "acceptable", "good", and "very good"
Oral acceptability | From pretreatment (month 0) until month 6 of the 6-month treatment period
  Evaluation of the oral acceptability on a 100mm VAS (from 0mm - very easy to swallow to 100mm - very difficult to swallow) of the treatment at each visit
Tolerance: Number of related adverse events during the study | Throughout the 6-month treatment period
  Number of related adverse events during the study
Efficacy: Investigator's global satisfaction at each visit | From pretreatment (month 0) until month 6 of the 6-month treatment period
  Evaluation of the investigator's global satisfaction at each visit on a four level scale of "bad", "acceptable", "good", and "very good"

CONTACTS AND LOCATIONS:
Overall Officials: Marcio Steinbruch, MD, Principal Investigator — Hospital Albert Einstein; Renato Kaufman, MD, Principal Investigator — Universidade Estadual do Rio de Janeiro
Locations (1):
- Centro Universitário Serra dos Órgãos - UNIFESO, Teresópolis, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No